CLINICAL TRIAL: NCT05653622
Title: Simultaneous Integrated Boost FDOPA PET Guided in Patients With Partially- or Non-operated Glioblastoma
Brief Title: Simultaneous Integrated Boost FDOPA Positron Emission Tomography (PET) Guided in Patients With Partially- or Non-operated Glioblastoma
Acronym: SIB-DOPA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Paul Strauss (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-010
Record Dates: First submitted 2022-11-28; First posted 2022-12-16 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Glioblastoma Multiforme, Adult
Keywords: glioblastoma; intensity modulated radiation therapy; 18F-DOPA-PET imaging
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SIB-DOPA (Experimental)
  Interventions: Procedure: Integrated boost technique (SIB) guided by PET FDOPA

INTERVENTIONS:
Procedure: Integrated boost technique (SIB) guided by PET FDOPA — intensity-modulated irradiation scheme with integrated boost technique (SIB) guided by PET FDOPA during the chemo-radiotherapy

SUMMARY:
Glioblastoma (GBM) is the most common primary brain cancer in adults. Surgery, chemoradiotherapy (temozolomide TMZ) and then adjuvant TMZ is the standard treatment. But, most patients relapse in a median time of 8-9 months; the median overall survival (OS) ranged from 15 to 18 months.

Some frail patients received hypofractionated radiation and concomitant and adjuvant TMZ. For some, the radiation dose is not optimal. Moreover, recurrences develop mainly in the initial tumor site. These two reasons justify increasing the dose. To limit the movements of these fragile patients, the method consists of increasing the dose without increasing the number of sessions by using the Simultaneous Integrated Boost (SIB) which increases the dose in targeted volumes while the rest of the volume receives a minimum dose. A phase I trial showed the possibility of increasing the dose in SIB up to 80 Gy in a part of the GBM enhanced on MRI.

FDOPA PET detects certain more aggressive tumor areas, areas likely to recur. Integrating them into the SIB seems appropriate. A phase II trial showed the interest of SIB guided by FDOPA PET in terms of progression-free survival but without impact on OS. This study differed from the one the investigators propose, because a dose and conventional fractionation, identical to that of the European Organization for Research and Treatment of Cancer/National Cancer Information Center (NCIC/EORTC) protocol were delivered, the gliomas were unmethylated MGMT, less likely to respond. Studies with SIB and hypofractionation are often retrospective and for others, hypofractionation was debatable and the dose increase was not based on PET capture but on MRI. However, a prospective phase II study, with SIB and hypofractionation, not integrating FDopa PET has demonstrated the relevance of SIB.

In this project, the investigators propose to use the integrated boost technique (SIB) guided by PET FDOPA to increase the radiation dose in GBM, in patients either fragile and partially operated, or only biopsied and for whom the prognosis is the most pejorative.

ELIGIBILITY:
Inclusion Criteria:

* Unfit patient without indication to the STUPP protocol :

Cohort 1 : Non-operable patients and ≥ 18 years old or ≤ 70 years old and Karnofsky Index (KI) ≥ 50% on inclusion AND Result of a biopsy available Cohort 2 : Patients > 70 years old and Balducci score I or II and KI ≥ 60% on inclusion AND Partial resection (defined on the remnographic criteria of postoperative MRI) OR biopsy result available

* Histologically proven glioblastoma
* Increased metabolism of amino acids in PET FDOPA allowing contouring the Biological Target Volume (BTV)

Exclusion Criteria:

* Patients with an indication for irradiation according to the STUPP protocol (fit patient)
* Patient with a contraindication to MRI or PET
* Limit of the provisional target volume or Planning target volume (PTV), second PTV < 2 cm from the chiasm and the optic nerves
* Absence of uptake of FDopa

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | At 24 months after inclusion
  Evaluate the overall survival (OS) of patients with glioblastoma treated with integrated boost (SIB) with increased dose guided by FDOPA PET

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | At 24 months after inclusion
  To assess the progression-free survival (PFS) of patients with glioblastoma treated with SIB with increased dose guided by FDOPA PET
Sites of progression: distant, marginal or in-field progression | At the date of progression, assessed up to 24 months
  The progression will be defined by its location by comparing the progression imaging with that used for dosimetry. It will be considered "distant" if it develops beyond the 95% isodose, "marginal" if it cuts the 95% isodose and "in-field" if it is completely within the 95% isodose. The 95% isodose is the reference isodose for the prescription of hypofractionated radiotherapy.
Assess the rate of acute complications of grade ≥ 3 | At 6 months after the start of radiotherapy
  Acute toxicities are defined as toxicities by the Common Terminology Criteria for Adverse Events (CTCAE v5) occurring within 6 months of the start of radiotherapy.
Characterize the PET parameters during progression | At the date of progression, assessed up to 24 months
  PET Parameters:
  * Standardized Uptake Value (SUV) max tumor, SUV max tumor/healthy tissue, SUV max T/striatum
  * SUV mean tumor, SUV mean tumor/healthy tissue, SUV mean T/striatum
Evolution of the PET parameters | Change between baseline and the date of progression, assessed up to 24 months
  PET Parameters:
  * Standardized Uptake Value (SUV) max tumor, SUV max tumor/healthy tissue, SUV max T/striatum
  * SUV mean tumor, SUV mean tumor/healthy tissue, SUV mean T/striatum
Assess quality of life measured with Quality of Life Questionnaire-Cancer 30items (QLQ-C30) | At inclusion
  The quality of life will be measured at the inclusion with Quality of Life Questionnaire-C30 (Cancer 30items).
  All items are scored 1 (worse outcome) to 4 (better outcome) or 1 (worse outcome) to 7 (better outcome). All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Assess quality of life measured with Quality of Life Questionnaire-Brain Neoplasms 20items (QLQ-BN20) | At inclusion
  The quality of life will be measured at the inclusion with Quality of Life Questionnaire - BN20 (Brain Neoplasms 20items).
  All items are scored 1 (worse outcome) to 4 (better outcome). All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Assess quality of life measured with Quality of Life Questionnaire-Cancer 30items (QLQ-C30) | At 3 months after inclusion
  The quality of life will be measured at 3 months with Quality of Life Questionnaire-C30 (Cancer 30items).
  All items are scored 1 (worse outcome) to 4 (better outcome) or 1 (worse outcome) to 7 (better outcome). All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Assess quality of life measured with Quality of Life Questionnaire-Brain Neoplasms 20items (QLQ-BN20) | At 3 months after inclusion
  The quality of life will be measured at 3 months with Quality of Life Questionnaire - BN20 (Brain Neoplasms 20items).
  All items are scored 1 (worse outcome) to 4 (better outcome). All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Assess quality of life measured with Quality of Life Questionnaire-Cancer 30items (QLQ-C30) | At 6 months after inclusion
  The quality of life will be measured at 6 months with Quality of Life Questionnaire-C30 (Cancer 30items).
  All items are scored 1 (worse outcome) to 4 (better outcome) or 1 (worse outcome) to 7 (better outcome). All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Assess quality of life measured with Quality of Life Questionnaire-Brain Neoplasms 20items (QLQ-BN20) | At 6 months after inclusion
  The quality of life will be measured at 6 months with Quality of Life Questionnaire - BN20 (Brain Neoplasms 20items).
  All items are scored 1 (worse outcome) to 4 (better outcome). All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Assess quality of life measured with Quality of Life Questionnaire-Cancer 30items (QLQ-C30) | At 12 months after inclusion
  The quality of life will be measured at 12 months with Quality of Life Questionnaire-C30 (Cancer 30items).
  All items are scored 1 (worse outcome) to 4 (better outcome) or 1 (worse outcome) to 7 (better outcome). All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Assess quality of life measured with Quality of Life Questionnaire-Brain Neoplasms 20items (QLQ-BN20) | At 12 months after inclusion
  The quality of life will be measured at 12 months with Quality of Life Questionnaire - BN20 (Brain Neoplasms 20items).
  All items are scored 1 (worse outcome) to 4 (better outcome). All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Assess quality of life measured with Quality of Life Questionnaire-Cancer 30items (QLQ-C30) | At 18 months after inclusion
  The quality of life will be measured at 18 months with Quality of Life Questionnaire-C30 (Cancer 30items).
  All items are scored 1 (worse outcome) to 4 (better outcome) or 1 (worse outcome) to 7 (better outcome). All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Assess quality of life measured with Quality of Life Questionnaire-Brain Neoplasms 20items (QLQ-BN20) | At 18 months after inclusion
  The quality of life will be measured at 18 months with Quality of Life Questionnaire - BN20 (Brain Neoplasms 20items).
  All items are scored 1 (worse outcome) to 4 (better outcome). All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Correlate O6-Methylguanine-DNA Methyltransferase (MGMT) promoter methylation status and Overall survival | At 24 months after inclusion
  MGMT promoter methylation status (binary variable, determined by either Polymerase Chain reaction (PCR) or immunohistochemistry)
Correlate O6-Methylguanine-DNA Methyltransferase (MGMT) promoter methylation status and Progression-Free Survival | At 24 months after inclusion
  MGMT promoter methylation status (binary variable, determined by either PCR or immunohistochemistry)
Correlate O6-Methylguanine-DNA Methyltransferase (MGMT) promoter methylation status and acute toxicities | At 24 months after inclusion
  MGMT promoter methylation status (binary variable, determined by either PCR or immunohistochemistry)

CONTACTS AND LOCATIONS:
Overall Officials: Caroline BUND, Principal Investigator — Centre Paul Strauss
Locations (3):
- France (3):
  - CHRU de Nancy, Nancy, De
  - Centre Paul Strauss, Strasbourg
  - ICL, Vandœuvre-lès-Nancy

REFERENCES:
- [Background] Perry JR, Laperriere N, O'Callaghan CJ, Brandes AA, Menten J, Phillips C, Fay M, Nishikawa R, Cairncross JG, Roa W, Osoba D, Rossiter JP, Sahgal A, Hirte H, Laigle-Donadey F, Franceschi E, Chinot O, Golfinopoulos V, Fariselli L, Wick A, Feuvret L, Back M, Tills M, Winch C, Baumert BG, Wick W, Ding K, Mason WP; Trial Investigators. Short-Course Radiation plus Temozolomide in Elderly Patients with Glioblastoma. N Engl J Med. 2017 Mar 16;376(11):1027-1037. doi: 10.1056/NEJMoa1611977. PMID 28296618
- [Background] Truc G, Bernier V, Mirjolet C, Dalban C, Mazoyer F, Bonnetain F, Blanchard N, Lagneau E, Maingon P, Noel G. A phase I dose escalation study using simultaneous integrated-boost IMRT with temozolomide in patients with unifocal glioblastoma. Cancer Radiother. 2016 May;20(3):193-8. doi: 10.1016/j.canrad.2015.12.005. Epub 2016 Apr 23. PMID 27117900
- [Background] Somme F, Bender L, Namer IJ, Noel G, Bund C. Usefulness of 18F-FDOPA PET for the management of primary brain tumors: a systematic review of the literature. Cancer Imaging. 2020 Oct 6;20(1):70. doi: 10.1186/s40644-020-00348-5. PMID 33023662